CLINICAL TRIAL: NCT04305392
Title: Pharmacokinetics, Pharmacodynamics and Safety of SHR4640 in Patients With Hepatic Impairment (Multicenter, Single Dose, Parallel, Open)
Brief Title: Pharmacokinetics, Pharmacodynamics and Safety of SHR4640 in Patients With Hepatic Impairment
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR4640-105
Record Dates: First submitted 2020-03-10; First posted 2020-03-12 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — ruzinurad

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal liver function (Experimental): Patients will receive single dose of SHR4640
  Interventions: Drug: SHR4640
- Mild Hepatic Impairment (Experimental): Patients will receive single dose of SHR4640
  Interventions: Drug: SHR4640
- Moderate Hepatic Impairment (Experimental): Patients will receive single dose of SHR4640
  Interventions: Drug: SHR4640

INTERVENTIONS:
Drug: SHR4640 — orally SHR4640

SUMMARY:
Study to evaluate pharmacokinetics, pharmacodynamics and safety of SHR4640 in patients with mild, moderate hepatic impairment and normal liver function in phase I clinical study.

ELIGIBILITY:
Inclusion Criteria:

-

All subjects:

* Signing the informed consent forms.
* 18 years to 65 years (inclusive).
* Body mass index should be between 18 and 30 kg/m2 (inclusive).
* No medication was used before screening#or stable medication for 4 weeks.

Normal liver function:

• Clinical laboratory tests during the screening period were normal or the abnormality has no clinical significance.

Hepatic impaired subjects:

* Child-Pugh Classification score clinically determined as mild or moderate hepatic impairment.
* Liver damage due to primary liver disease.

Exclusion Criteria:

-

All subjects:

• Subject known or suspected of being sensitive to the study drugs or its ingredient.

Normal liver function:

* Previous history of liver function impairment, or physical examination and laboratory examination at screening indicated the presence or possibility of liver function impairment.
* Hepatitis B surface antigen (HBsAg) positive or Anti-hepatitis C virus (HCV) antibody or hepatitis C core antigen positive within 3 months prior to administration.

Hepatic impaired subjects:

* Suspected or diagnosed as liver cancer or with other malignant tumors.
* Drug induced liver injury#acute liver injury#liver transplantation history.
* Subjects with hepatic failure,or severe complications caused by Hepatocirrhosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 72 hours after dosing
  Peak Plasma Concentration (Cmax) will be compared between normal hepatic function patients and mild or moderate hepatic dysfunction patients
Area under the plasma concentration versus time curve from single dosing time extrapolated to infinity (AUC0-∞) | 72 hours after dosing
  Area under the plasma concentration versus time curve from single dosing time extrapolated to infinity (AUC0-∞) will be compared between normal hepatic function patients and mild or moderate hepatic dysfunction patients

CONTACTS AND LOCATIONS:
Locations (1):
- Meixia Wang, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided